CLINICAL TRIAL: NCT00184964
Title: The Validation of Coregistered CT-PET Imaging in Determining Tumor Volume and Atelectasis in Patients With Operable Non-Small-Cell Lung Cancer and Tumor Associated Atelectasis With Histological Examination of the Resected Specimen
Brief Title: Validation of Coregistered CT-PET Imaging in Determining Tumor Volume and Atelectasis in Patients With Operable Non-Small-Cell Lung Cancer and Tumor Associated Atelectasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004/032
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Carcinoma, Non Small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: CT-scan, PET-scan

SUMMARY:
CT-PET image fusion has the potential to differentiate 'tumor' from 'atelectasis' much better than the CT-scan in patients with non-small cell lung cancer who also have atelectasis.

This however has never been validated on a histological level. In this study patients with non small cell lung cancer and atelectasis who are eligible for surgery undergo a CT-scan and a PET-scan prior to surgery.

The resection specimen will be compared to the preoperative imaging.

ELIGIBILITY:
Inclusion Criteria:

-Patients with non small cell lung cancer and atelectasis, who are eligible for surgery.

Exclusion Criteria:

* age < 18 years
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2004-06

PRIMARY OUTCOMES:
Histological validation of CT-PET image fusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bussink, MD, PhD, Study Director — Radiation oncologist, Radboud University Nijmegen Medical Centre, Nijmegen, The Netherlands
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands